CLINICAL TRIAL: NCT01953549
Title: Physical Fitness Training in Subacute Stroke (PHYS-Stroke)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Agnes Flöel, Prof. Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHYS-Stroke
Record Dates: First submitted 2013-06-28; First posted 2013-10-01 (Estimated); Last update posted 2019-06-06 (Actual); Status verified 2019-06

CONDITIONS: Stroke
Keywords: physical activity, relaxation, activities of daily living, motor functions, cognitive functions
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- physical fitness training (Experimental): aerobic physical fitness training
  Interventions: Procedure: physical fitness training
- relaxation (Active Comparator): non-aerobic training
  Interventions: Procedure: relaxation

INTERVENTIONS:
Procedure: physical fitness training
  Arms: physical fitness training
Procedure: relaxation
  Arms: relaxation

SUMMARY:
The aim of this study is to investigate whether a 4-week physical fitness training (target intervention) in stroke patients (subacute stage) increase the walking speed and activities of daily living compared with a control intervention (relaxation exercises). The target or control intervention is performed in addition to standard rehabilitation treatment.

ELIGIBILITY:
Inclusion Criteria for patients:

* diagnosis of stroke within 5-45 days after stroke
* age >= 18 years
* able to sit for at least 30 seconds
* Barthel index < =65 at inclusion
* considered able to perform aerobic exercise as determined by responsible physician
* Written informed consent of the patient

Exclusion Criteria:

* Patient considered unable to comply with study requirements
* stroke due to intracranial hemorrhage primarily due to bleeding from ruptured aneurysm or arteriovenous malformation
* patients with progressive stroke
* unable to perfom the required exercises due to

  1. medical problems
  2. musculo-skeletal problems
  3. neurological problems
* required help to at least 1 persons to walk before stroke due to neurological or non-neurological co-morbidities
* life expectancy of less than 1 year as determined by responsible physician
* alcohol or drug addiction within the last 6 months
* significant current psychiatric illness as defined as medication-refractory of bipolar affective disorder, psychosis, schizophrenia or suicidality
* current participation in another intervention study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-10; Primary Completion 2017-07-06 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Gait speed and Barthel Index (BI) (co-primary endpoint) | 3 months post stroke vs baseline
  comparing gait speed (m/s) and points achieved in BARTHEL Index in aerobic and non-aroebic training group 3 months after stroke vs baseline (before intervention)

SECONDARY OUTCOMES:
Gait speed and Barthel Index (BI) | directly after intervention; 6 months post stroke; all vs baseline
  comparing gait speed (m/s) and points achieved in BI in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 6 months post stroke vs baseline (before intervention)
motor function | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing motor function (assessed via different clinical scales e.g. Rivermead Arm test, REPAS, Box and Block Test, Medical Research Council Scale) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
mobility | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing different mobilitiy indices like gait endurance (in min), stride length, step cadence, use of walking aids, actigraph measurements and the Rivermead mobility Index in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
cognitive function | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing cognitive function (assessed via points achieved in different scales, e.g. Montreal Cognitive Assessment, Trail Making test, word fluency) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
Disability | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing disability (Modified rankin scale) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
Quality of life (QoL) | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing QoL (EQ-5D-5L scale) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
sleep | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing sleep quality (Pittsburgh sleep quality index) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
mood | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing mood (CES-D scale) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
Physical fitness | directly after intervention; 3 months post stroke; 6 months post stroke, all vs baseline
  comparing gait energy Expenditure in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
Assessment of safety | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing different criteria (recurrent fatal or non-fatal cardiovascular or cerebrovascular events, refferal to acute hospital, death) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention)
Maximal walking speed and Barthel-Index | 3 months post stroke vs. baseline
  per Protocol analysis of co-primary endpoint (pre-specified in statistical analysis plan and protocol)

OTHER OUTCOMES:
resting systolic and diastolic blood pressure | directly after intervention; 3 months post stroke; 6 months post stroke, all vs baseline
  comparing resting systolic and diastolic blood pressure (mmHg) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
laboratory parameters | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing different laboratory parameters (derived by blood draw) like hormones, hemogram, liver and kidney function, and coagulation parameters in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
hair cortisol concentration | at baseline
  hair cortisol concentration by taking a small strand of hair is measured at baseline; part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
resting heart rate | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comaparing resting heart rate(beats/minute) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
waist to hip ratio | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing waist to hip ratio (cm) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
markers of peripheral immunity | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comapring markers of peripheral immunity (e.g., monocytic HLA-DR expression) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
lipid profile | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing lipide such as triglycerides, cholesterol (total, LDL,HDL, and LP(a)) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
blood glucose | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing insulin, glucose, and HbA1c in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
markers of inflammation | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing markers of inflammation (e.g., including Interleukin (IL) 6, 1b, hs-CRP) in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
body mass index | directly after intervention; 3 months post stroke; 6 months post stroke; all vs baseline
  comparing body mass index in aerobic and non-aroebic training group after the 4-week intervention interval as well as after 3 and after 6 months post stroke vs baseline (before intervention); part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
Endothelial function | directly after intervention vs. baseline
  the endothelial function of included patients will be assessed prospectively before and after the 4 week intervention with the Endopat2000 device. First measurement was conducted in January 11th 2014. Results will be correlated with imaging and blood-derived biomarkers as well as differences between intervention groups; part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)
Magnetic resonance imaging parameters | directly after intervention vs. baseline
  Primary and secondary endpoints are specified after completion of the interim analysis after inclusion of the first 24 patients (first stage). In a second stage the study is conducted with specified primary and secondary endpoints with recruitment of up to 76 remaining patients; part of substudy 'Biomarkers and Perfusion - Training-Induced Changes After Stroke (BAPTISe)' - NCT01954797 (will be analyzed seperately)

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (7):
  - Beelitz Heilstätten, Beelitz-Heilstätten, Brandenburg
  - Median Klinik Grünheide, Grünheide, Brandenburg
  - Charité - Universitätsmedizin Berlin, Berlin
  - Charité Campus Benjamin Franklin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Evanglisches Geriatriezentrum Berlin, Berlin
  - Medical Park Berlin, Berlin

REFERENCES:
- [Background] Floel A, Werner C, Grittner U, Hesse S, Jobges M, Knauss J, Seifert M, Steinhagen-Thiessen E, Govercin M, Dohle C, Fischer W, Schlieder R, Nave AH, Meisel A, Ebinger M, Wellwood I. Physical fitness training in Subacute Stroke (PHYS-STROKE)--study protocol for a randomised controlled trial. Trials. 2014 Feb 3;15:45. doi: 10.1186/1745-6215-15-45. PMID 24491065
- [Derived] Rackoll T, Hinrichs T, Neumann K, Wolfarth B, Nave AH; Phys-Stroke Study Group. Improvements in Walking During Subacute Stroke Rehabilitation Translate to Physical Activity at the Chronic Stage: A Sub-Analysis From the Phys Stroke Trial. Brain Neurorehabil. 2024 Oct 28;17(3):e17. doi: 10.12786/bn.2024.17.e17. eCollection 2024 Nov. PMID 39649709
- [Derived] Kirzinger B, Stroux A, Rackoll T, Endres M, Floel A, Ebinger M, Nave AH. Elevated Serum Inflammatory Markers in Subacute Stroke Are Associated With Clinical Outcome but Not Modified by Aerobic Fitness Training: Results of the Randomized Controlled PHYS-STROKE Trial. Front Neurol. 2021 Aug 26;12:713018. doi: 10.3389/fneur.2021.713018. eCollection 2021. PMID 34512526
- [Derived] Nave AH, Rackoll T, Grittner U, Blasing H, Gorsler A, Nabavi DG, Audebert HJ, Klostermann F, Muller-Werdan U, Steinhagen-Thiessen E, Meisel A, Endres M, Hesse S, Ebinger M, Floel A. Physical Fitness Training in Patients with Subacute Stroke (PHYS-STROKE): multicentre, randomised controlled, endpoint blinded trial. BMJ. 2019 Sep 18;366:l5101. doi: 10.1136/bmj.l5101. PMID 31533934
- Available data/document: Statistical Analysis Plan — https://doi.org/10.6084/m9.figshare.5375026.v1 — Statistical Analysis Plan of PHYS-Stroke Trial. If download path is offline please contact torsten.rackoll@charite.de

DOCUMENTS (1):
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT01953549/SAP_000.pdf